CLINICAL TRIAL: NCT06778278
Title: Adapting Behavioral Activation to Improve Mental Health Outcomes and Reduce Suicide Risk During the Military Transition
Brief Title: Transition Health and Resilience Through Valued Experiences (THRiVE) Pilot for Newly Separated Veterans
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RTI International (Other)
Collaborators: U.S. Army Medical Research Acquisition Activity (U.S. Federal Agency)
Responsible Party: Principal Investigator, Shannon Blakey, Research Clinical Psychologist, RTI International
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0219706; HT94252410947 (Other Grant/Funding Number: Assistant Secretary of Defense for Health Affairs endorsed by the Department of Defense); CDMRP-TP230060 (Other: Assistant Secretary of Defense for Health Affairs endorsed by the Department of Defense); 24-08-666-907 (Other: Biomedical Research Alliance of New York)
Record Dates: First submitted 2025-01-09; First posted 2025-01-16 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Military Transition; Community Reintegration; Mental Health; Suicidal Ideation; Alcohol Misuse
Keywords: Military transition; Community reintegration; Mental health; Suicidal ideation; Transitioning Service Members; Newly separated Veterans
MeSH Terms: conditions — Psychological Well-Being; Suicidal Ideation | interventions — Health Transition; Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- THRiVE (Experimental)
  Interventions: Behavioral: Transition Health and Resilience through Valued Experiences (THRiVE) Program

INTERVENTIONS:
Behavioral: Transition Health and Resilience through Valued Experiences (THRiVE) Program — Six (6) total weekly, 90-minute, small-group, peer-led sessions delivered virtually

SUMMARY:
The objective of this study is to develop and pilot a program designed to improve mental health outcomes and reduce suicide risk during the transition from military to civilian life. It is hypothesized that the Transition Health and Resilience through Valued Experiences (THRiVE) program, to be developed as part of this study, will meet participant recruitment, retention, and satisfaction benchmarks (primary outcomes) and show positive preliminary effects on mental health symptoms, risk factors for suicidal ideation, and psychosocial functioning outcomes (secondary outcomes).

The specific aims of this study are to:

1. Develop a small-group, peer-led, cross-cutting prevention program for newly separated veterans (NSVs) called THRiVE and
2. Evaluate the feasibility, acceptability, and preliminary effects of the THRiVE program on mental health symptoms, risk factors for suicidal ideation, and psychosocial functioning outcomes.

Up to 40 NSVs participating in this Stage 1 pilot study will complete validated self-report measures at baseline, immediately after completing the THRiVE program (post-THRiVE), and 3 months after completing the THRiVE program (follow-up). The duration of a participant's time in the study is anticipated to be 5 months.

DETAILED DESCRIPTION:
Transition from military to civilian life presents both opportunities and challenges. Although existing programs provide newly separated veterans (NSVs) with valuable support for their vocational well-being during the military transition, these programs do not fully address the psychosocial aspects of reintegrating into civilian life. This is problematic because the military transition is a time during which NSVs are at higher risk for developing mental health disorders and suicidal ideation. Although evidence-based treatments for common mental health concerns exist, cross-cutting prevention programs for NSVs are lacking. Behavioral Activation (BA), an evidence-based treatment that holds potential for optimizing psychosocial well-being during the military transition, could be adapted into a skills-based mental health promotion and suicide prevention program to fill this gap. This Phase 1 study involves a one-arm clinical trial to pilot test the program, called Transition Health and Resilience through Valued Experiences (THRiVE), in a sample of up to 40 NSVs. Primary outcomes include measures of feasibility (based on administrative data) and acceptability (based on administrative data and a validated self-report instrument). Mental health symptoms, risk factors for suicidal ideation, and psychosocial functioning will be assessed (using validated self-report instruments) at baseline, immediately post-THRiVE, and at follow-up 3 months after completing the THRiVE program. The duration of a participant's time in the study is anticipated to be 5 months. Findings from this pilot study will inform the design an anticipated larger, fully powered Stage 2 trial.

ELIGIBILITY:
Inclusion Criteria:

* Be a United States military veteran
* Have separated/retired from the military no more than 12 months prior to study enrollment
* Be at least 18 years old
* Have access to the internet; a desktop computer, laptop, tablet, or other "smart" device with video camera, speakers, and microphone; and a private place from which to attend THRiVE sessions
* Reside and complete all study activities within the United States

Exclusion Criteria:

* Endorse lifetime manic, hypomanic, or psychotic episodes
* Meet Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria for current severe alcohol use disorder or substance use disorder (except for tobacco use disorder, which will not be exclusionary)
* Screen positive for moderate or high acute risk for suicide
* Screen positive for more than minimal risk for other-directed violence
* Are receiving or plan to receive BA therapy for any mental health condition between enrollment and the 3-month follow-up assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Participant recruitment rate | 14 months
  The percentage of NSVs who are determined to be eligible based on their eligibility assessment and choose to enroll. It is anticipated that recruitment will begin May 2025 and enrollment of the final participant will be July 2026 (a recruitment/enrollment window of 14 months).
Participant retention rate | Through completion of the THRiVE group, an average of 2 months
  The percentage of participants who attend at least 4 of the 6 planned total THRiVE sessions
Client Satisfaction Questionnaire-8 | At completion of the THRiVE group, an average of 2 months
  Participant self-reported satisfaction with the THRiVE program at post-THRiVE. Possible scale scores range 8 to 32, with higher scores indicating greater program satisfaction.

SECONDARY OUTCOMES:
Generalized Anxiety Disorder-7 | Through study completion, an average of 5 months
  Changes in past-2-week anxiety symptoms from baseline to follow-up. Possible scale scores range 0 to 21, with higher scores indicating greater anxiety symptom severity.
PTSD Checklist for DSM-5 | Through study completion, an average of 5 months
  Changes in past-month posttraumatic stress symptoms from baseline to follow-up. Possible scale scores range 0 to 80, with higher scores indicating greater posttraumatic stress symptom severity.
Alcohol Use Disorders Identification Test | Through study completion, an average of 5 months
  Changes in hazardous or harmful alcohol use from baseline to follow-up. Possible scale scores range 0 to 40, with higher scores indicating more hazardous or harmful alcohol use.
Drug Abuse Screening Test | Through study completion, an average of 5 months
  Changes in drug misuse consequences from baseline to follow-up. Possible scale scores range 0 to 10, with higher scores indicating greater drug misuse consequences.
Patient Health Questionnaire-9 | Through study completion, an average of 5 months
  Changes in past-2-week depression symptoms from baseline to follow-up. Possible scale scores range 0 to 27, with higher scores indicating greater depression symptom severity.
Interpersonal Needs Questionnaire | Through study completion, an average of 5 months
  Changes in thwarted belongingness and perceived burdensomeness from baseline to follow-up. Possible thwarted belongingness subscale scores range 9 to 63, with higher scores indicating greater thwarted belongingness. Possible perceived burdensomeness subscale scores range 6 to 42, with higher scores indicating greater perceived burdensomeness.
Positive and Negative Suicide Ideation Inventory | Through study completion, an average of 5 months
  Changes in past-2-week protective and negative risk dimensions of suicidal ideation from baseline to follow-up. Possible protective dimension subscale scores range 6 to 30, with higher scores indicating greater protective factors. Possible negative risk dimension subscale scores range 8 to 40, with higher scores indicating greater negative risk factors.
Military to Civilian Questionnaire | Through study completion, an average of 5 months
  Changes in psychosocial functioning from baseline to follow-up. Possible scale scores range 0 to 4, with higher scores indicating greater difficulties with psychosocial functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon M Blakey, PhD, Principal Investigator — RTI International
Locations (1):
- RTI International, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Blakey SM, Vandermaas-Peeler JR, Counts J, Croxford J, Rae Olmsted KL, Gant P, Elbogen EB, Asman K. Bringing veteran mental health promotion and suicide prevention efforts upstream: The THRiVE study protocol. Contemp Clin Trials. 2025 Nov;158:108100. doi: 10.1016/j.cct.2025.108100. Epub 2025 Oct 4. PMID 41052716